CLINICAL TRIAL: NCT03840603
Title: PROARRAY : Impact on PCT+ FilmArray RP2 Plus Use in LRTI Suspicion in Emergency Department
Brief Title: Impact on PCT+ FilmArray RP2 Plus Use in LRTI Suspicion in Emergency Department
Acronym: PROARRAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioMérieux (Industry)
Collaborators: APHP (Other); BioFortis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2018-A02173-52
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Tract Infections
Keywords: Respiratory Tract Infections; Emergency Department; Procalcitonin
MeSH Terms: conditions — Respiratory Tract Infections; Emergencies

STUDY DESIGN:
Intervention Model Description: This is an open label, prospective, single-center, randomized interventional trial with 2 arms (FilmArray-guided arm versus usual care).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Usual care of patients with suspected Low RespiratoryTract Infection at the discretion of the attending physician. Care may entail a CRP and/or a PCT measurement, but no nasopharyngeal swab sampling.
- Film Array RP2 Assay guided (Experimental): In the emergency room a nasopharyngeal swab sample will be collected from subjects with a suspected Low RespiratoryTract Infection for the Film Array RP2 Assay guided plus a blood sample for the PCT assay if the PCT measurement has not been already prescribed.
  Interventions: Diagnostic Test: Film Array RP2 Assay guided

INTERVENTIONS:
Diagnostic Test: Film Array RP2 Assay guided — Nasopharyngeal swab sample collected from subjects with a suspected LRTI for the Film Array RP2 assay plus a blood sample for the PCT assay.
  Arms: Film Array RP2 Assay guided

SUMMARY:
The real-time reporting of PCT results along with viral PCR data from the FilmArray® Respiratory Panel 2 plus in conjunction with an antimicrobial stewardship plan will aid in the proper withholding or withdrawing of antibiotics (ATB) when the collective data is indicative of a viral Lower Respiratory Tract Infection (LRTI).

The addition of the FilmArray® RP2plus diagnostic test indicating the presence of a viral infection in subjects presenting with respiratory symptoms could improve the confidence to care-providing physicians to withhold prescribing antibiotics.

DETAILED DESCRIPTION:
In the emergency room a nasopharyngeal swab sample will be collected from subjects with a suspected LRTI for the FilmArray respiratory panel assay plus a blood sample for the PCT assay if the PCT measurement has not been already prescribed.

The FilmArray® Respiratory Panel 2 plus (RP2plus) is a multiplexed nucleic acid test intended for use with FilmArray® 2.0 or FilmArray® Torch systems for the simultaneous qualitative detection and identification of multiple respiratory viral and bacterial nucleic acids in nasopharyngeal swabs (NPS) obtained from individuals suspected of respiratory tract infections.

Both results will be reported in real-time to the treating physicians with the recommendation to withhold or withdraw antibiotics if:

1. PCT<0.10 µg/L with either a positive (with a viral respiratory pathogen) or negative FilmArray assay or
2. PCT<0.25 µg/L and FilmArray positive with a viral respiratory pathogen. For the control arm, patients will benefit from the usual care of patients with suspected LRTI at the discretion of the attending physician. Care may entail a CRP and/or a PCT measurement, but no nasopharyngeal swab sampling.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject is ≥ 18 years of age attending the ED with LRTI symptom defined as at least one among:

  1. sweats, chills, body aches and pain, temperature >38°C) and at least one among:
  2. cough, sputum production, dyspnea, chest pain, altered breath sounds at auscultation.
* 2. Subject signs informed consent

Exclusion Criteria:

1. Subject is a prisoner
2. Subject is a Pregnant
3. Subject has no social insurance
4. Subject is enrolled in end of life care
5. Subject refuses to participate in study procedures
6. Subject is already enrolled (each patient will only be tested one time with the FilmArray® RP2plus)
7. Subject has a contraindication (per the discretion of the attending physician) to a nasopharyngeal swab (for example, nose bone fracture or recent history of maxilla-facial surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Duration of total antibiotic exposure | First 28 days
  The primary endpoint in this study is the duration of total antibiotic exposure (measured in days) in the first 28 days after randomization.

SECONDARY OUTCOMES:
Initiation of an antibiotic therapy | First 28 days
  initiation of an antibiotic therapy in the first 28 days after the reporting test results to clinicians (both ATB given in the ED or given a prescription for an ATB to get at the pharmacy)
Protocol "failure" within 15 days of randomization | within 15 days
  protocol "failure" within 15 days of randomization (defined as worsening of LRTI and/or receipt of antibiotics in cases where no initial ATB treatment was administered, and/or unplanned ED's re-admission for the same complaint)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Hausfater, Principal Investigator — Hôpital Pitié-Salpêtrière, APHP
Locations (1):
- AP-HP Pitié la salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albrich WC, Dusemund F, Bucher B, Meyer S, Thomann R, Kuhn F, Bassetti S, Sprenger M, Bachli E, Sigrist T, Schwietert M, Amin D, Hausfater P, Carre E, Gaillat J, Schuetz P, Regez K, Bossart R, Schild U, Mueller B; ProREAL Study Team. Effectiveness and safety of procalcitonin-guided antibiotic therapy in lower respiratory tract infections in "real life": an international, multicenter poststudy survey (ProREAL). Arch Intern Med. 2012 May 14;172(9):715-22. doi: 10.1001/archinternmed.2012.770. PMID 22782201
- [Background] Branche AR, Walsh EE, Vargas R, Hulbert B, Formica MA, Baran A, Peterson DR, Falsey AR. Serum Procalcitonin Measurement and Viral Testing to Guide Antibiotic Use for Respiratory Infections in Hospitalized Adults: A Randomized Controlled Trial. J Infect Dis. 2015 Dec 1;212(11):1692-700. doi: 10.1093/infdis/jiv252. Epub 2015 Apr 24. PMID 25910632
- [Background] Das D, Le Floch H, Houhou N, Epelboin L, Hausfater P, Khalil A, Ray P, Duval X, Claessens YE, Leport C; ESCAPED Study Group. Viruses detected by systematic multiplex polymerase chain reaction in adults with suspected community-acquired pneumonia attending emergency departments in France. Clin Microbiol Infect. 2015 Jun;21(6):608.e1-8. doi: 10.1016/j.cmi.2015.02.014. Epub 2015 Feb 20. PMID 25704448
- [Background] Woodhead M, Blasi F, Ewig S, Garau J, Huchon G, Ieven M, Ortqvist A, Schaberg T, Torres A, van der Heijden G, Read R, Verheij TJ; Joint Taskforce of the European Respiratory Society and European Society for Clinical Microbiology and Infectious Diseases. Guidelines for the management of adult lower respiratory tract infections--full version. Clin Microbiol Infect. 2011 Nov;17 Suppl 6(Suppl 6):E1-59. doi: 10.1111/j.1469-0691.2011.03672.x. PMID 21951385